CLINICAL TRIAL: NCT02100774
Title: Effect of Genetic Variants of Intestinal Transporters of Lipophilic Micronutrients (Vitamins D, E and Carotenoids) on Absorption Efficiency of These Compounds.
Brief Title: Effect of Genetic Variants on Fat-soluble Vitamin Bioavailability
Acronym: VITAGENES
Status: Completed | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Marseille (Other)
Responsible Party: Principal Investigator, Patrick Borel, INRAE Research Director, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Other Study IDs: 2008-A00955-50
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2014-03

CONDITIONS: Biological Availability of Vitamins and Micronutrients
Keywords: bioavailability; postprandial period; genetic variants; single nucleotide polymorphisms; vitamin; carotenoid; lutein; lycopene; tocopherol; cholecalciferol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood, adipose tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- healthy male adults: no added micronutrient, tomato puree, lutein supplement, vitamin E supplement, vitamin D supplement

SUMMARY:
The aim was to identify minor genetic variations (single nucleotide polymorphisms) that explain the interindividual variability in bioavailability of fat soluble micronutrients (fat soluble vitamins and carotenoids).

DETAILED DESCRIPTION:
Healthy male volunteers were genotyped and submitted to 5 test-meals containing either no micronutrient of interest, 100 g tomato puree as a source of carotenoids, a lutein supplement, a vitamin E supplement or a vitamin D supplement. Blood samples were taken in the postprandial period (up to 8 hours after the test-meals intake) and the concentration of the studied micronutrients were measured in the chylomicrons. Multivariate analysis were then performed to identify single nucleotide polymorphisms that best explained the variance in the interindividual response (0 to 8 h area under the curve) in micronutrients.

ELIGIBILITY:
Inclusion Criteria:

gender : male age : 18 to 60 years old BMI: [18 to 29.9] kg/m2 Fasting Cholesterol concentration : < 2,5 g/l Fasting triglyceride concentration < 2 g/l Fasting glycemia ≤ 1,1 g/l Fasting Hemoglobin < 13 g/dl HIV as well as hepatitis C and B negative

Exclusion Criteria:

smokers regular consumption of vitamin supplement > 140 g/week alcohol vegetarian diseases drugs assumed to affect the metabolism of lipids or fat soluble micronutrients (e.g. ezetimibe)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy male adults.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
micronutrient concentration in plasma chylomicrons | 8 hours
  The subjects were submitted to test-meals rich in micronutrients of interest and the ability of each subject to absorb the studied micronutrients was evaluated by measuring the postprandial chylomicron response (0 to 8 h area under the curve of the chylomicron micronutrient concentration) in each micronutrient.

SECONDARY OUTCOMES:
micronutrient concentration in adipose tissue | 8 hours
  A first sample of adipose tissue was taken before the intake of the test-meal rich in fat soluble micronutrients. A second sample was taken 8 h after the test-meal intake. The aim was to assess whether the consumption of the studied fat soluble micronutrient modified the concentration of this micronutrient in adipose tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Borel, PhD, Study Director — INRA/INSERM/Aix-Marseille University
Locations (1):
- Centre d'Investigation Clinique de l'hôpital de la Conception, Marseille, France

REFERENCES:
- [Background] Borel P. Genetic variations involved in interindividual variability in carotenoid status. Mol Nutr Food Res. 2012 Feb;56(2):228-40. doi: 10.1002/mnfr.201100322. Epub 2011 Sep 29. PMID 21957063
- [Derived] Zumaraga MP, Desmarchelier C, Gleize B, Nowicki M, Ould-Ali D, Landrier JF, Borel P. Identification of Genetic Polymorphisms Associated with Interindividual Variability of Vitamin A Concentration in Adipose Tissue of Healthy Male Adults. J Nutr. 2024 Dec;154(12):3693-3703. doi: 10.1016/j.tjnut.2024.10.035. Epub 2024 Oct 21. PMID 39442757
- [Derived] Zumaraga MP, Desmarchelier C, Gleize B, Nowicki M, Ould-Ali D, Borel P. Characterization of the interindividual variability of lutein and zeaxanthin concentrations in the adipose tissue of healthy male adults and identification of combinations of genetic variants associated with it. Food Funct. 2024 Sep 30;15(19):9995-10006. doi: 10.1039/d4fo03087g. PMID 39279719
- [Derived] Desmarchelier C, Borel P, Goncalves A, Kopec R, Nowicki M, Morange S, Lesavre N, Portugal H, Reboul E. A Combination of Single-Nucleotide Polymorphisms Is Associated with Interindividual Variability in Cholecalciferol Bioavailability in Healthy Men. J Nutr. 2016 Dec;146(12):2421-2428. doi: 10.3945/jn.116.237115. Epub 2016 Oct 26. PMID 27798339
- [Derived] Borel P, Desmarchelier C, Nowicki M, Bott R. A Combination of Single-Nucleotide Polymorphisms Is Associated with Interindividual Variability in Dietary beta-Carotene Bioavailability in Healthy Men. J Nutr. 2015 Aug;145(8):1740-7. doi: 10.3945/jn.115.212837. Epub 2015 Jun 10. PMID 26063065
- [Derived] Borel P, Desmarchelier C, Nowicki M, Bott R, Morange S, Lesavre N. Interindividual variability of lutein bioavailability in healthy men: characterization, genetic variants involved, and relation with fasting plasma lutein concentration. Am J Clin Nutr. 2014 Jul;100(1):168-75. doi: 10.3945/ajcn.114.085720. Epub 2014 May 7. PMID 24808487